CLINICAL TRIAL: NCT04645459
Title: The Influence of Low Phosphorus Meals on Serum Phosphorus Concentration and Inflammatory Indicators in Hemodialysis Patients
Brief Title: The Influence of Low Phosphorus in Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: N202004062
Record Dates: First submitted 2020-10-15; First posted 2020-11-27 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-05

CONDITIONS: Hemodialysis Patients

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low phosphorus meal group (LP group) (Experimental): The proteins of the low phosphorus meal had been removed by an average 20 -30% of the phosphorus through boiling the meats before cooking process.
  Interventions: Other: low phosphorus meals
- control group (Placebo Comparator): The boiling method did not process for the control meals.
  Interventions: Other: control meals

INTERVENTIONS:
Other: low phosphorus meals — All subjects followed their usual diets but took one tablet of calcium carbonate as phosphate binder per meal for the first week washout diet. After washout diet, subjects were assign to control or study group randomly and entered to the study period for one week. The diets of the study group were low phosphorus ( LP group), but the dietary phosphorous levels of the control group were not modified. During the study period, all subjects including LP group and control group still kept their usually accustomed behavior about regular breakfast and also took one tablet of calcium carbonate as phosphate binder with every breakfast meal. The LP group and control group replaced daily lunch and dinner with low phosphorus and standard meals respectively and should not take any phosphate binder during the study period for one week.
  Arms: low phosphorus meal group (LP group)
Other: control meals — All subjects followed their usual diets but took one tablet of calcium carbonate as phosphate binder per meal for the first week washout diet. After washout diet, subjects were assign to control or study group randomly and entered to the study period for one week. The diets of the study group were low phosphorus ( LP group), but the dietary phosphorous levels of the control group were not modified. During the study period, all subjects including LP group and control group still kept their usually accustomed behavior about regular breakfast and also took one tablet of calcium carbonate as phosphate binder with every breakfast meal. The LP group and control group replaced daily lunch and dinner with low phosphorus and standard meals respectively and should not take any phosphate binder during the study period for one week.
  Arms: control group

SUMMARY:
Consuming high levels of dietary phosphate and poor adherence of phosphate-binding-therapy might induce hyperphosphatemia in the hemodialysis (HD) patients. Therefore, the risks of Chronic Kidney Disease-related Mineral and Bone Disorders (CKD-MBDs) and inflammation will be increased. This double blind and intervention randomized controlled trial study will be designed to investigate the hypothesis that if low phosphorus meals decrease serum phosphorus concentration and inflammatory indicators. A total of 80 HD patients in the HD center of Shuang Ho Hospital will be recruited and be assigned to low phosphorus meal group (LP group) and control group randomly before one-week-washout period. The subjects of LP group and control group will consume low phosphorus meals and standard meals respectively. During washout period and study period, all subjects will continue to consume their regular breakfast and take one tablet of calcium carbonate with meal. All data will be collected at baseline, one week after the washout period, and the end of the 7-days-study period. The indicators are including dietary contents, phosphate binder administration, indicators of dialysis adequacy, nutritional indicators, blood lipid indicators, biochemical indicators, CKD-MBDs indicators, and inflammation indicators. Data were analyzed by Statistical Product and Service Solutions program version 18. Paired t-test, Student's t-test, Pearson correlation coefficient and Logistic regression will be used. P < 0.05 will be considered as statistically significant.

DETAILED DESCRIPTION:
Study Design and Subjects:

This study was design as a randomized, double-blind control trail. A total of 80 HD patients were recruited from the HD center of Taipei Medical University-Shuang Ho Hospital in Taiwan. The inclusion criteria were including ≧20 years old and non vegetarian. The exclusion criteria are including liver dysfunction, cancer and pregnancy.

Dietary Intervention:

All subjects followed their usual diets but took one tablet of calcium carbonate as phosphate binder per meal for the first week washout diet. After washout diet, subjects were assign to control or study group randomly and entered to the study period for one week. The diets of the study group were low phosphorus ( LP group), but the dietary phosphorous levels of the control group were not modified. During the study period, all subjects including LP group and control group still kept their usually accustomed behavior about regular breakfast and also took one tablet of calcium carbonate as phosphate binder with every breakfast meal. The LP group and control group replaced daily lunch and dinner with low phosphorus and standard meals respectively and should not take any phosphate binder during the study period for one week.

For controlling the volumes of proteins, phosphorus and calcium easily, the main courses of both of the study and the control meals were made by a central kitchen. All of the meals contained 3 exchanges of protein (25 g) and 1 exchange of vegetable. There were 5 main courses for the both diets. The proteins of the study meals had been removed by an average 20 -30% of the phosphorus through boiling the meats before cooking process. But the boiling method did not process for the control meals. Every meal including all the study and the control meals contained one tablet of calcium carbonate. As a consequence, the additional phosphate binders should not be taken while eating the study meals. The subjects had to prepare carbohydrate by themselves, and they could choose any source of carbohydrate as their wants.

Data Collection:

The personal characteristics and the anthropometry data were collected at baseline. All data were collected at baseline, one week after the washout period, and the end of the 7-days-study period. The indicators were including dietary contents, phosphate binder administration, dialysis adequacy, nutritional indicators, blood lipid indicators, biochemical indicators, CKD-MBDs indicators, and inflammation indicators.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients, ≥ 20 years of age

Exclusion Criteria:

* ≥ 80 years of age, liver cirrhosis, cancer, pregnancy, vegetarian

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-12-03 (Estimated); Primary Completion 2021-05-28 (Estimated); Study Completion 2021-05-28 (Estimated)

PRIMARY OUTCOMES:
anthropometric measurement | baseline
  body height (cm)
anthropometric measurement | one week after the washout period
  body height (cm)
anthropometric measurement | the end of the 7-days-study period
  body height (cm)
anthropometric measurement | baseline
  body weight before hemodialysis (Kg), dry weight (Kg)
anthropometric measurement | one week after the washout period
  body weight before hemodialysis (Kg), dry weight (Kg)
anthropometric measurement | the end of the 7-days-study period
  body weight before hemodialysis (Kg), dry weight (Kg)
blood pressure | baseline
  systolic blood pressure (mmHg), diastolic blood pressure (mmHg)
blood pressure | one week after the washout period
  systolic blood pressure (mmHg), diastolic blood pressure (mmHg)
blood pressure | the end of the 7-days-study period
  systolic blood pressure (mmHg), diastolic blood pressure (mmHg)
dietary contents | baseline
  24-hour dietary recall
dietary contents | one week after the washout period
  24-hour dietary recall
dietary contents | the end of the 7-days-study period
  24-hour dietary recall
phosphate binder administration | baseline
  type and dosing frequency
phosphate binder administration | one week after the washout period
  type and dosing frequency
phosphate binder administration | the end of the 7-days-study period
  type and dosing frequency
indicators of dialysis adequacy | baseline
  Kt/V
indicators of dialysis adequacy | one week after the washout period
  Kt/V
indicators of dialysis adequacy | the end of the 7-days-study period
  Kt/V
blood lipid indicators | baseline
  LDL(mg/dL), HDL (mg/dL) , cholesterol (mg/dL) , triglyceride (mg/dL)
blood lipid indicators | one week after the washout period
  LDL(mg/dL), HDL (mg/dL) , cholesterol (mg/dL) , triglyceride (mg/dL)
blood lipid indicators | the end of the 7-days-study period
  LDL(mg/dL), HDL (mg/dL) , cholesterol (mg/dL) , triglyceride (mg/dL)
biochemical indicators | baseline
  normalized protein equivalent of total nitrogen appearance(g/kg/d)
biochemical indicators | one week after the washout period
  normalized protein equivalent of total nitrogen appearance(g/kg/d)
biochemical indicators | the end of the 7-days-study period
  normalized protein equivalent of total nitrogen appearance(g/kg/d)
biochemical indicators | baseline
  pre-Alb(mg/dL)
biochemical indicators | one week after the washout period
  pre-Alb(mg/dL)
biochemical indicators | the end of the 7-days-study period
  pre-Alb(mg/dL)
biochemical indicators | baseline
  ferritin(ng/mL)
biochemical indicators | one week after the washout period
  ferritin(ng/mL)
biochemical indicators | the end of the 7-days-study period
  ferritin(ng/mL)
biochemical indicators | baseline
  red blood cell (10^6/μL), white blood count(10^3/μL)
biochemical indicators | one week after the washout period
  red blood cell (10^6/μL), white blood count(10^3/μL)
biochemical indicators | the end of the 7-days-study period
  red blood cell (10^6/μL), white blood count(10^3/μL)
biochemical indicators | baseline
  Hb (g/dL)
biochemical indicators | one week after the washout period
  Hb (g/dL)
biochemical indicators | the end of the 7-days-study period
  Hb (g/dL)
biochemical indicators | baseline
  Hct (%)
biochemical indicators | one week after the washout period
  Hct (%)
biochemical indicators | the end of the 7-days-study period
  Hct (%)
biochemical indicators | baseline
  FGF23
biochemical indicators | one week after the washout period
  FGF23
biochemical indicators | the end of the 7-days-study period
  FGF23
biochemical indicators | baseline
  iPTH (pg/mL)
biochemical indicators | one week after the washout period
  iPTH (pg/mL)
biochemical indicators | the end of the 7-days-study period
  iPTH (pg/mL)
biochemical indicators | baseline
  blood urea nitrogen(mg/dL) , creatinine(mg/dL) , uric acid(mg/dL)
biochemical indicators | one week after the washout period
  blood urea nitrogen(mg/dL) , creatinine(mg/dL) , uric acid(mg/dL)
biochemical indicators | the end of the 7-days-study period
  blood urea nitrogen(mg/dL) , creatinine(mg/dL) , uric acid(mg/dL)
biochemical indicators | baseline
  estimated glomerular filtration rate (ml/min/1.73m^2)
biochemical indicators | one week after the washout period
  estimated glomerular filtration rate (ml/min/1.73m^2)
biochemical indicators | the end of the 7-days-study period
  estimated glomerular filtration rate (ml/min/1.73m^2)
inflammation indicators | baseline
  C reactive protein (mg/dL)
inflammation indicators | one week after the washout period
  C reactive protein (mg/dL)
inflammation indicators | the end of the 7-days-study period
  C reactive protein (mg/dL)
inflammation indicators | baseline
  interleukin-1 (pg/mL) , interleukin-6 (pg/mL) , tumor necrosis factor-α (pg/mL)
inflammation indicators | one week after the washout period
  interleukin-1 (pg/mL) , interleukin-6 (pg/mL) , tumor necrosis factor-α (pg/mL)
inflammation indicators | the end of the 7-days-study period
  interleukin-1 (pg/mL) , interleukin-6 (pg/mL) , tumor necrosis factor-α (pg/mL)
Electrolyte | baseline
  P(mg/dL), Ca(mg/dL), Mg(mg/dL)
Electrolyte | one week after the washout period
  P(mg/dL), Ca(mg/dL), Mg(mg/dL)
Electrolyte | the end of the 7-days-study period
  P(mg/dL), Ca(mg/dL), Mg(mg/dL)
Electrolyte | baseline
  K(mEq/L), Na(mEq/L)
Electrolyte | one week after the washout period
  K(mEq/L), Na(mEq/L)
Electrolyte | the end of the 7-days-study period
  K(mEq/L), Na(mEq/L)

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Szu Wu, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No